CLINICAL TRIAL: NCT04037579
Title: Protocol for a Non-randomized Survey to Evaluate Social Skills and Physical Capacity Improvement in Down Syndrome People Who Routinely Practice Sports. Self and Observers´ Perception.
Brief Title: Protocol for a Non-randomized Survey in Down Syndrome People Who Practice Sports. Self and Observers´ Perception.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Estrella Agüera Buendía, Professor. Responsible of AGR-019 Research Group, Universidad de Córdoba
Other Study IDs: University of Cordoba, Spain
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Down Syndrome; Social Skills; Physical Activity
Keywords: physical activity; self-determination; Social inclusion; Well-being; Rights; Interpersonal relations
MeSH Terms: conditions — Down Syndrome; Social Skills; Motor Activity; Social Inclusion | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Down Syndrome Cordoba Association: The participant will answer a questionnaire related to social skills and physical activity
  Interventions: Other: Survey
- Down Syndrome Granada Association: The participant will answer a questionnaire related to social skills and physical activity
  Interventions: Other: Survey
- Down Syndrome Malaga Association: The participant will answer a questionnaire related to social skills and physical activity
  Interventions: Other: Survey
- Observers in Cordoba: Observers from Cordoba, Spain who know Down Syndrome people well (at least for six months) will answer a questionnaire related to their social skills and physical activity
  Interventions: Other: Survey
- Observers in Granada: Observers from Granada, Spain who know Down Syndrome people well (at least for six months) will answer a questionnaire related to their social skills and physical activity
  Interventions: Other: Survey
- Observers in Malaga: Observers from Malaga, Spain who know Down Syndrome people well (at least for six months) will answer a questionnaire related to their social skills and physical activity
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Non-randomised survey

SUMMARY:
This survey arises from one objective of a PhD thesis whose purpose is to "Identify what social skills people with Down syndrome have that do a routine activity and compare them with those developed by those SD people who perform sports activities."

DETAILED DESCRIPTION:
This study is a non-randomized survey. The aim of the current protocol is to describe how will be the process to get information about the participant, the questionnaire design and how was validated and the planned analysis of results.

Participants: Around 150 Down Syndrome people from Cordoba, Malaga y Granada who belong to The Down Syndrome association and 150 parents, family, tutors, teachers etc.

Consent process: Before designing the survey, consent was requested from the management team Down of Córdoba, Malaga and Gradana associations, as well as family members, parents, tutors, teachers, etc.

Standard Operating Procedures: First, RC (author) gathered as much information as possible about the subject under study and selected the most important topics related to the research focus. After that, the questionnaire was designed modifying the KidsLife-Down Scale. The questionnaire will be divided into three parts.

An introduction to the questionnaire describes the instructions, structure, the reasons for the study and confidentiality in accordance with the Spanish Organic Law 3/2018 on the Protection.

The first part of the questionnaire will assess self-perception from people with Down about their social skills. The second will evaluate the opinion of this issue from other people who know them well (at least for six months) and who have the opportunity to observe the person evaluated for extended periods of time (parents, family, tutors, teachers etc.). Finally, for the third part, it will be used the International Physical Activity Questionnaire (IPAQ) for the purpose of collecting information about the types of physical activity do in their daily routines. The questions will be referred to the time they have been physically active in the last 7 days.

Second, the questionnaire was sent to the Down Syndrome Association of Córdoba (DSAC) so that they reviewed the possible mistakes made when defining the questions and validate it. After that, Down Malaga and Down Granada Association found the questionnaire understandable and acceptable.

Third, they gave the corresponding feedback that served to formulate the questions in the appropriate way to avoid confusion in the surveyed.

The questionnaire will be sent by e-mail to the Cordoba Association and a paper version will available for participants. From Córdoba, it will be spread to Málaga and Granada Associations in order it will be distributed among associates.

Analysis of results: Estimated outcomes will be percentages of agreement with each answer. Data from all surveys will be analyzed. The statistical study will be carried out with the SPSS 24.0 program. The mean value and standard deviation (± SD) of each item will be calculated on a numerical scale. Statistical analysis will be performed with parametric tests, t-Student for related samples. The level of statistical significance will be calculated.

Two of the authors (RC and JC) will analyse de data, and results will be discussed among the work team.

Conducting a pilot test or pre-test before applying the survey will help to detect possible failures and optimize the results of our survey. Despite its importance, should not consider the pilot study as a substitute for a careful wording of the questionnaire.

Report on the survey: Before writing the report, It will be reviewed the data for errors and inconsistencies. Make sure the data reflects exactly what the survey concludes. The conclusion will summarize the results.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome
* Do sport
* Belonging to Cordoba, Mágala and Granada Associatio

Exclusion Criteria:

* Others metal incapacities
* Others Asociation

Ages: 10 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Down Syndrome people who practise sports and a people who know them well (at least for six months) and who have the opportunity to observe person evaluated for extended periods of time (parents, family, tutors, teachers etc.).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-26 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Sport effect on social skills in Down Syndrome people | 6 months
  To Evaluate sport effect on social skills in Down Syndrome people using a survey

SECONDARY OUTCOMES:
Types of physical activities carried out by Down Syndrome people | 6 months
  To know which types of physical activities are carried out by Down Syndrome people using a survey

CONTACTS AND LOCATIONS:
Overall Officials: Estrella Agüera, Dotor, Study Director — Universidad de Córdoba
Locations (1):
- Estrella Agüera, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access request will be reviewed by an external Independent Review Panel. Requestors will be required to sing a Data Access Agreement.